CLINICAL TRIAL: NCT03481127
Title: Implementation and Evaluation of Psychological Services Integration in Gynecological Oncology Clinics
Brief Title: Psychological Services Integration in Gynecological Oncology Clinics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201711117
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Gynecologic Oncology Patient
MeSH Terms: interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Usual Care (Active Comparator): -No psychosocial care in clinic
  Interventions: Other: Surveys; Procedure: Blood draw; Procedure: Fresh tissue from ovary
- Arm 2: Integrated Care (Experimental): -Those who receive integrated care will receive a one-page care plan completed by Dr. Vanderlan including their scores from screening questionnaires , recommendations for coping strategies and available supportive resources.
  Interventions: Behavioral: Integrated psychological care; Other: Surveys; Procedure: Blood draw; Procedure: Fresh tissue from ovary

INTERVENTIONS:
Behavioral: Integrated psychological care — Additional possible strategies used may include supportive or validating interventions, increasing/introducing/reinforcing coping strategies, psychoeducation; distress tolerance skills; brief cognitive behavioral therapy; cognitive restructuring; activity scheduling; acceptance; and relaxation/mindfulness.
  Arms: Arm 2: Integrated Care
Other: Surveys — * NCCN Distress Thermometer
  * PROMIS Depression & Anxiety
  * Quality of Life (SF-12)
  * Brief COPE
  * Patient awareness and satisfaction survey
Procedure: Blood draw — * For patients with ovarian, fallopian tube, or primary peritoneal cysts
  * Optional
  * Enrollment, 3 months after enrollment, and 6 months after enrollment
Procedure: Fresh tissue from ovary — * For patients with ovarian, fallopian tube, or primary peritoneal cysts
  * Optional
  * At time of standard of care surgery

SUMMARY:
The purpose of this study is to understand the feasibility and impact of integrated psychological care in outpatient gynecologic oncology clinics with the goal of creating a new standard of care. The investigators propose an intervention study comparing patient-centered outcomes (assessed by surveys) between women who receive usual care versus integrated psychological care. The investigators' objectives are to learn about the process of integration of psychological care directly into outpatient gynecologic oncology clinics and the impact of such integration on patients' well-being, presentation of symptoms, psychological functioning, coping mechanisms, awareness of support services offered, and perception of quality of care. As this is a feasibility study, aims are focused on assessing patient willingness for psychological intervention in the medical office, provider willingness to have psychologist present in clinic, and impact of psychological intervention. With such data to warrant further integration and time of psychologists in medical clinics, next steps for immediate and long-term projects may include focus on high risk populations, specific disease sites, additional provider clinics, more psychologist time spent in gynecological oncology clinics, and effectiveness of interventions with higher power. The investigators hope the results will serve as preliminary data for an integrated psychosocial care model that can be implemented in other oncology clinics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Scheduled for an appointment in a gynecologic oncology clinic at the Siteman Cancer Center at the Center for Advanced Medicine or the Women's Tumor Clinic at the Center for Outpatient Health at Barnes-Jewish Hospital
* Patients may or may not have a cancer diagnosis.
* All gynecologic cancer types, histologic grades, primary or recurrent disease.
* Patients actively undergoing treatment or close observation
* Pregnant or lactating patients
* Able to speak and read English
* Able to consent

Inclusion criteria (correlative studies only) -Patients who are undergoing pre-operative work-up for evaluation of an adnexal mass by a Washington University gynecologic oncologist.

Exclusion Criteria:

-Impaired by a psychiatric or cognitive disorder that limits their ability to give consent or communicate with their medical providers about symptoms (as determined by the patient's medical team)

Exclusion criteria (correlative studies only)

* Neoadjuvant chemotherapy
* Treatment within the past month with antidepressant medications that affect serotonin physiology
* Specific histology: low malignant potential tumors, non-epithelial cancer histology.
* Previous cancer diagnosis within the past five years or recurrent cancer
* Regular steroid use in the last month
* Presence of comorbidities with known effects on the immune system (e.g., systemic lupus erythematosus, multiple sclerosis, and rheumatoid arthritis), congestive heart failure, pregnancy, or stroke within the past six months
* Major surgery in the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of integrating psychosocial care by a trained psychologist into gynecologic cancer outpatient clinics as measured by patient enrollment | Completion of patient enrollment (approximately 12 months)
  -Willingness to participate with integrated care as quantified by proportion of enrolled patients from the number of approached eligible patients

SECONDARY OUTCOMES:
Provider willingness to have a psychologist present | 6 months after start of study enrollment
  -5 item survey about willingness to have psychologist present in clinic
Differences in clinic visit duration with and without a psychologist present | Day 1
  -Clinic visit duration is defined as the time from check-in to patient discharge
Difference in psychological correlates of daily functioning as measured by patient distress between women who receive usual care versus integrated psychological care | Enrollment, 3 months after enrollment, and 6 months after enrollment
  * NCCN Distress Thermometer: picture of thermometer that states to circle the number that best describes how much distress has been experienced in the past week (10=extreme distress and 0=no distress)
  * Next section contains categories of Practical Problems, Family Problems, Emotional Problems, Physical Problems, Spiritual/religious concerns - participant is to mark yes or no to indicate if they have had problems in the past week
  * The distress thermometer score of 0-10 is recorded. The problem areas endorsements are tallied within each problem area.
Difference in psychological correlates of daily functioning as measured by patient depression between women who receive usual care versus integrated psychological care | Enrollment, 3 months after enrollment, and 6 months after enrollment
  * PROMIS Depression & Anxiety - asks participant in the last 7 days if they have felt worthless, helpless, depressed, hopeless, fearful, lack of focus, worrying, and uneasy. Check box choices are never, rarely, sometimes, often, and always
  * Each question has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. Never = 1, rarely = 2, sometimes = 3, often =4, always = 5. Points are added to raw score. Raw score is converted to t-score via short form conversion table.
Difference in psychological correlates of daily functioning as measured by patient anxiety between women who receive usual care versus integrated psychological care | Enrollment, 3 months after enrollment, and 6 months after enrollment
  * PROMIS Depression & Anxiety - asks participant in the last 7 days if they have felt worthless, helpless, depressed, hopeless, fearful, lack of focus, worrying, and uneasy. Check box choices are never, rarely, sometimes, often, and always
  * Point values are as follows: never =1, rarely, rarely = 2, sometimes = 3, often =4, always = 5. Points are added to raw score. Raw score is converted to t-score via short form conversion table.
Difference in psychological correlates of daily functioning as measured by patient quality of life between women who receive usual care versus integrated psychological care | Enrollment, 3 months after enrollment, and 6 months after enrollment
  * Quality of life (SF-12): 12 item survey
  * Scores are recoded to give numerical value, with some items reverse scored. Scoring is broken down into mental health and physical health subscale scores.
Difference in psychological correlates of daily functioning as measured by patient coping mechanisms between women who receive usual care versus integrated psychological care | Enrollment, 3 months after enrollment, and 6 months after enrollment
  * Brief COPE: 28 item survey with answers ranging from 1=I haven't been doing this at all to 4=I've been doing this a lot
  * Scores are on tallied based on answers to 4 point likert scale. No reverse scoring. There are 14 subscales with two questions each.
Difference in psychological correlates of perception of psychological care as measured by patient perception of Siteman Cancer Center being highly focused on their wellbeing between women who receive usual care versus integrated psychological care | Enrollment, 3 months after enrollment, and 6 months after enrollment
  * 4 item survey
  * Each question has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question.
  * 1=strongly disagree to 5=strongly agree
Difference in psychological correlates of awareness of psychological care as measured by awareness of support services offered between women who receive usual care versus integrated psychological care | Enrollment, 3 months after enrollment, and 6 months after enrollment
  * 4 item survey
  * Each question has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question.
    * 1=strongly disagree to 5=strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Vanderlan, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu